CLINICAL TRIAL: NCT05011604
Title: Full-Digital Workflow in Single-Tooth Implant Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francesco Gianfreda (Other)
Responsible Party: Sponsor-Investigator, Francesco Gianfreda, PhD Student, University of Rome Tor Vergata
Organization: University of Rome Tor Vergata (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180171
Record Dates: First submitted 2021-08-07; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Full Digital Workflow; Edentulous Jaw; Implant Site Reaction
Keywords: Full-Digital Workflow; Single-Tooth Implant Rehabilitation; Digital Dentistry
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: A total of 19 patients (22 implants) were included in the present study with mean follow-up time of 2 years. A full-digital workflow was performed on each patient through the design and printing of a surgical guide, the taking of the impression with an intraoral scanner and the CAD-CAM design of the crowns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implant Failure (Other): Early peri-implantitis and failed osseointegration.
  Interventions: Device: Full-Digital Workflow in Single-Tooth Implant Rehabilitation

INTERVENTIONS:
Device: Full-Digital Workflow in Single-Tooth Implant Rehabilitation — For all patients included in the study, a digital impression was taken using an intraoral scanner. A CBCT exam was performed on the mandibular or maxillary jaw with the missing tooth. The stl. and the dicom. files were then superimposed to allow the surgical planning.
  Then it was elevated and reflected to increase the volume on the buccal side and exposed the bone surface. After this point, the implant was inserted, and another digital impression was taken.
  Sutures 6.0 were positioned after healing abutment positioning to stabilize the soft tissues.
  The final abutment and the provisional were designed and manufactured using cad-cam technology. One week thereafter, definitive abutment was positioned. Provisional restoration was then cemented using provisional cement removing all the possible occlusal contacts both in protrusive and in lateral positions. Three months thereafter, once osteointegration was obtained, definitive zirconia restoration was positioned and cemented.

SUMMARY:
The digital workflow in dental implantology has been used for planning the cases with the intraoral scanners and computer tomography, together helping clinicians to be more accurate and precise. Today, thanks to digital technology clinicians can plan from surgical to the final prosthesis using 3D models and cad-cam machines. The aim of this research is to validate the full digital workflow for the single-tooth implant rehabilitation. A total of 19 patients (22 implants) were included in the present study with mean follow-up time of 2 years. A full-digital workflow was performed on each patient through the design and printing of a surgical guide, the taking of the impression with an intraoral scanner and the CAD-CAM design of the crowns.

DETAILED DESCRIPTION:
Study design The present study was a retrospective case series conducted in one clinical center in accordance with the Good Clinical Practice Guidelines (GCPs) following the recommendations of the World Medical Association Declaration of Helsinki-ethical principles for medical research involving human subjects as revised in Fortaleza (2013).

All patients were informed about the benefits and the possible risks of a fully digital workflow and its alternatives finally a signed written consent was obtained. Subject population

The current retrospective study was performed in a private clinic in Rome, Italy, where all patients treated by the same operator between January 2017 and June 2020 were consecutively enrolled:

* Patients older than 18 years
* Patients in good health (Asa 1 or Asa 2)
* Patients with healthy periodontium (probing pocket depth ≤ 4 mm, no bleeding on probing)
* Patients not requiring bone augmentation procedures Patients requiring a single implant supported reconstructions were included in the present study.

Surgical and prosthetic workflow For all patients included in the study, a digital impression was taken using an intraoral scanner (CS3600, Carestream Dental, Atlanta, Ga). During the same day, a CBCT (CS9000 3D, Carestream Dental, Atlanta, Ga) exam was performed on the mandibular or maxillary jaw with the missing tooth. The stl. and the dicom. files were then superimposed to allow the surgical planning (RealGuide, 3Diemme, Cantù, Italy).

One week after planning, implant insertion was performed after the elevation of a flap with a papilla preservation technique. Once designed, the flap was dis-epitelized using a diamond bur. Then it was elevated and reflected to increase the volume on the buccal side and exposed the bone surface. After this point, the implant (Sweden & Martina, Padua, Italy) was inserted, and another digital impression was taken.

Sutures 6.0 were positioned (monofilament-polyglecaprone suture, Surgiclryl-Monofast ®SMI-Belgium) after healing abutment positioning to stabilize the soft tissues.

In the mean, time, the file of the impression was sent to technician and the final abutment and the provisional were designed and manufactured using cad-cam technology. One week thereafter, definitive abutment was positioned and screwed at 25N/cm Provisional restoration was then cemented using provisional cement (Temp Bond, Kerr Sybron Dental Specialities, Washington, DC, USA) removing all the possible occlusal contacts both in protrusive and in lateral positions.

Sutures were removed 2 weeks postoperative. Three months thereafter, once osteointegration was obtained, definitive zirconia restoration was positioned and cemented.

Eventual deficiencies of the prosthetic rehabilitation at the time of provisional restoration (contact points, esthetics) were noticed and fixed directly adding composite. In all these cases, a new impression after soft tissue maturation was performed and strategically, a new crown in PMMA was designed and realized. Final check before producing the zirconia element was performed positioning the crown on the abutment.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients in good health (Asa 1 or Asa 2)
* Patients with healthy periodontium (probing pocket depth ≤ 4 mm, no bleeding on probing)

Exclusion Criteria:

* Patients requiring bone augmentation procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Predictability in cases of intercalated edentulism | 1 year
  Implant success

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Canullo, Dentistry, Principal Investigator — Private Practice
Locations (1):
- Luigi Canullo, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
Individual patient data will be available on private request to the principal investigator

REFERENCES:
- [Background] da Silva Salomao GV, Chun EP, Panegaci RDS, Santos FT. Analysis of Digital Workflow in Implantology. Case Rep Dent. 2021 Feb 15;2021:6655908. doi: 10.1155/2021/6655908. eCollection 2021. PMID 33628525
- [Background] Stanley M, Paz AG, Miguel I, Coachman C. Fully digital workflow, integrating dental scan, smile design and CAD-CAM: case report. BMC Oral Health. 2018 Aug 7;18(1):134. doi: 10.1186/s12903-018-0597-0. PMID 30086753
- [Background] Flugge T, Derksen W, Te Poel J, Hassan B, Nelson K, Wismeijer D. Registration of cone beam computed tomography data and intraoral surface scans - A prerequisite for guided implant surgery with CAD/CAM drilling guides. Clin Oral Implants Res. 2017 Sep;28(9):1113-1118. doi: 10.1111/clr.12925. Epub 2016 Jul 20. PMID 27440381
- [Background] Mangano FG, Admakin O, Bonacina M, Lerner H, Rutkunas V, Mangano C. Trueness of 12 intraoral scanners in the full-arch implant impression: a comparative in vitro study. BMC Oral Health. 2020 Sep 22;20(1):263. doi: 10.1186/s12903-020-01254-9. PMID 32962680